CLINICAL TRIAL: NCT01437657
Title: A Randomized, Double-blind, Parallel-group Study of the Safety and Efficacy of RO4917523 Versus Placebo, as Adjunctive Therapy in Patients With Major Depressive Disorder With Inadequate Response to Ongoing Antidepressant Treatment
Brief Title: MARIGOLD Study: A Study of RO4917523 Versus Placebo as Adjunctive Therapy in Patients With Major Depressive Disorder and an Inadequate Response to Ongoing Antidepressant Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP25620; 2011-001436-33 (EudraCT Number)
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Matching RO4917523 placebo orally daily, 6 weeks
  Interventions: Drug: Placebo
- RO4917523 0.5 mg (Experimental): 0.5 mg orally daily, 6 weeks
  Interventions: Drug: RO4917523 0.5 mg
- RO4917523 1.5 mg (Experimental): 1.5 mg orally daily, 6 weeks
  Interventions: Drug: RO4917523 1.5 mg

INTERVENTIONS:
Drug: Placebo — Matching RO4917523 placebo orally daily, 6 weeks
  Arms: Placebo
Drug: RO4917523 0.5 mg — 0.5 mg orally daily, 6 weeks
  Arms: RO4917523 0.5 mg
Drug: RO4917523 1.5 mg — 1.5 mg orally daily, 6 weeks
  Arms: RO4917523 1.5 mg

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group study will evaluate the safety and efficacy of RO4917523 as adjunctive therapy in patients with major depressive disorder and an inadequate response to ongoing antidepressant therapy. Anticipated time on study treatment is 6 weeks with a 3-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, 18 to 70 years of age at time of informed consent
* Major depressive disorder without psychotic features as defined by DSM-IV-TR criteria
* Inadequate response to ongoing antidepressant treatment, as defined by protocol
* Body mass index (BMI) 18 to 38 kg/m2 inclusive

Exclusion Criteria:

* Currently receiving treatment with a combination of antidepressants (two or more), or an adjunctive potentiating treatment as defined by protocol
* Previously received RO4917523
* History of failure, or utilization during the current episode of Electroconvulsive Therapy (ECT) or repetitive Transcranial Magnetic Stimulation (rTMS)
* History of use at any time of Vagus Nerve Stimulation (VNS) or Deep Brain Stimulation (DBS)
* Current or past history of bipolar disorder (e.g. manic, hypomanic, or mixed episodes)
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale (MADRS) | From baseline to Week 6

SECONDARY OUTCOMES:
Change in Clinical Global Impression Score - Severity (CGI-S) | From baseline to Week 6
Change in Clinical Global Impression Score - Improvement (CGI-I) | From baseline to Week 6
Safety: Incidence of adverse events | approximately 2 years
Proportion of patients exhibiting remission (MADRS </= 10) after 6 weeks of treatment | approximately 2 years
Proportion of patients exhibiting response (reduction in MADRS >/= 50% of baseline score) after 6 weeks of treatment | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (60):
- United States (25):
  - Little Rock, Arkansas
  - Costa Mesa, California
  - Garden Grove, California
  - Oceanside, California
  - Orange, California
  - Riverside, California
  - San Diego, California
  - Santa Ana, California
  - Wildomar, California
  - Atlanta, Georgia
  - Libertyville, Illinois
  - Naperville, Illinois
  - Oak Brook, Illinois
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Las Vegas, Nevada
  - Marlton, New Jersey
  - Brooklyn, New York
  - Cedarhurst, New York
  - Oklahoma City, Oklahoma
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Kirkland, Washington
- Chile (2):
  - Santiago
  - Temuco
- Germany (5):
  - Berlin
  - Freiburg im Breisgau
  - Hanover
  - Mainz
  - Wiesbaden
- Japan (10):
  - Chūōku
  - Hokkaido
  - Hyōgo
  - Kanagawa
  - Kita-ku
  - Kurayoshi-shi
  - Kyoto
  - Osaka
  - Shinjuku-ku
  - Tokyo
- Mexico (3):
  - Aguascalientes
  - León
  - Monterrey
- Poland (6):
  - Bełchatów
  - Bialystok
  - Choroszcz
  - Kielce
  - Lodz
  - Tuszyn
- Romania (5):
  - Bucharest
  - Constanța
  - Craiova
  - Targouiste
  - Târgu Mureş
- Saint Petersburg, Russia
- Taiwan (3):
  - Keelung
  - Taichung
  - Taipei

REFERENCES:
- [Derived] Quiroz JA, Tamburri P, Deptula D, Banken L, Beyer U, Rabbia M, Parkar N, Fontoura P, Santarelli L. Efficacy and Safety of Basimglurant as Adjunctive Therapy for Major Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jul 1;73(7):675-84. doi: 10.1001/jamapsychiatry.2016.0838. PMID 27304433